CLINICAL TRIAL: NCT05591014
Title: The Effectiveness of a Novel Software Program to Help in ROTEM Interpretation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Natalie Silverton, Associate Professor of Anesthesiology, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00159279
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Coagulation Disorder, Blood
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Intervention Model Description: The sensitivity/specificity and diagnostic accuracy of clinicians will be compared before and after the use of novel ROTEM app. The performance of more experienced clinicians will be compared to those with little to no experience in ROTEM. Analysis will be done using a mixed effects model to account for clustering of measurements within clinician groups. Inter-rater reliability analysis will be done to assess the similarity within clinician groups using the ICC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Software Tutorial (Experimental): Participants will be asked to interpret a series of ROTEM studies before and after a tutorial on a novel ROTEM interpretation software.
  Interventions: Device: Novel ROTEM interpretation software

INTERVENTIONS:
Device: Novel ROTEM interpretation software — Clinicians will be asked to interpret ROTEM studies before and after exposure to a novel ROTEM interpretation software.

SUMMARY:
The purpose of this study is to assess a novel rotational thromboelastometry (ROTEM®) interpretation software to determine whether its use improves the accuracy of clinician interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Current residents and attending physicians in the University of Utah Department of Anesthesiology who have a range of experience and exposure to thromboelastography

Exclusion Criteria:

* Refusal to consent or no longer an active member of the University of Utah Department of Anesthesiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 1 year of data collection
  sensitivity/specificity of clinician responses compared to a reference standard

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No